CLINICAL TRIAL: NCT00052559
Title: A Phase I Study Of The Antiangiogenic Agent Bevacizumab In Combination With 5-Fluourouracil And External Beam Radiation Therapy In Rectal Cancer
Brief Title: Bevacizumab, Fluorouracil, and External-Beam Radiation Therapy in Treating Patients With Stage II or Stage III Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02908; 6042-05-7R1; CDR0000258532; U01CA099118 (NIH); U01CA062490 (NIH)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Rectum; Stage II Rectal Cancer; Stage III Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil

ARMS (1):
- Treatment (bevacizumab, fluorouracil, radiation therapy) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 (courses 1-4). Beginning with course 2, patients also receive fluorouracil IV continuously on days 1-14 and undergo external beam radiotherapy on days 1-5 and 8-12. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Patients undergo surgery 7 weeks after completion of chemoradiotherapy.
  Cohorts of 6 patients receive escalating doses of bevacizumab until the MTD is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 20 additional patients are treated at the MTD.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Radiation: external beam radiation therapy; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Radiation: external beam radiation therapy — Undergo external beam radiation therapy
  Other Names: EBRT
Procedure: therapeutic conventional surgery — Undergo surgery
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of bevacizumab when given together with fluorouracil and external-beam radiation therapy in treating patients with stage II or stage III rectal cancer. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining monoclonal antibody therapy with chemotherapy and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of a vascular endothelial growth factor (VEGF) neutralizing antibody, bevacizumab, when administered concurrently with 5-fluorouracil (5-FU) and external beam radiation therapy (EBRT) in patients with clinical stage T3 or T4 rectal cancer prior to surgery.

II. To obtain preliminary data of the pathological response rate after preoperative therapy.

III. To obtain preliminary data regarding progression free survival, local control, and overall survival.

IV. To obtain preliminary data of the changes in the angiogenic profile of rectal cancer induced by this therapy.

OUTLINE: This is a multicenter, dose-escalation study of bevacizumab.

Patients receive bevacizumab IV over 30-90 minutes on day 1 (courses 1-4). Beginning with course 2, patients also receive fluorouracil IV continuously on days 1-14 and undergo external beam radiotherapy on days 1-5 and 8-12. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery 7 weeks after completion of chemoradiotherapy.

Cohorts of 6 patients receive escalating doses of bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 20 additional patients are treated at the MTD.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary adenocarcinoma of the rectum that begins within 15 cm of the anal verge as determined by sigmoidoscopy and/or colonoscopy
* Clinical T3 or T4 tumors as determined by the following features:

  * Tethered or fixed tumor on physical exam
  * cT3, cT4, or N+ disease must be confirmed by an endorectal ultrasound or surface coil MRI
* There must be no evidence of metastatic disease as confirmed by physical examination, chest radiograph, and abdominal/pelvic CT scan
* ECOG performance status 0, 1, 2 (Karnofsky >= 70%)
* Life expectancy of greater than 2 years
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of bevacizumab on the developing human fetus are unknown; for this reason and because radiation therapy and 5-FU agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients with no known HIV or HIV risk factors will be eligible for this study without HIV testing

Exclusion Criteria:

* Patients with a "concurrently active" second malignancy other than non- melanoma skin cancers or in situ cervical cancer are excluded; patients are not considered to have a "concurrently active" malignancy if they have completed therapy and considered by their physician to be at less than 30% risk of relapse at a minimum of 5 years after all therapy
* Prior Treatment:

  * No prior treatment for this malignancy
  * No prior history of pelvic irradiation
  * No prior history of 5-FU-based therapy for any malignancy
  * No prior treatment with bevacizumab
  * Patients must not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition bevacizumab or other agents used in study
* Bevacizumab - Specific exclusion criteria:

  * History or evidence upon physical examination of CNS disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke
  * Serious, non-healing wound, ulcer, or bone fracture
  * Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, history of myocardial infarction, unstable angina within 12 months), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 1 year prior to Day 0
  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; biopsies (other than rectal cancer) within 7 days prior to Day 0; placement of a vascular access device within 7 days prior to Day 0
  * Arterial thromboembolic events within previous 12 months including transient ischemic attack, cerebrovascular accident, unstable angina, myocardial infarction, or clinically significant peripheral vascular disease. Vascular surgery, stenting or angioplasty within previous 12 months; no history of venous thromboembolic events that require continuation of therapeutic dose of anticoagulation
  * Current or recent (within 10 days prior to Day 0) use of full-dose oral or parenteral anticoagulants or thrombolytic agents (except as required to maintain patency of preexisting, permanent indwelling IV catheters; for subjects receiving warfarin, international normalized ratio [INR] of < 1.5; appropriate use of heparin should be discussed with the Medical Monitor)
  * Chronic, daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti- inflammatory medications (of the kind known to inhibit platelet function at doses used to treat chronic inflammatory diseases)
  * Presence of bleeding diathesis or coagulopathy
  * Active infection requiring parenteral antibiotics on Day 0
  * Proteinuria at baseline or clinically significant impairment of renal function
  * Subjects unexpectedly discovered to have >= 1+ proteinuria during screening should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate < 1 gram protein/24 hr to allow participation in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because bevacizumab, radiation therapy, and 5-FU have potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bevacizumab, breastfeeding should be discontinued if the mother is treated with bevacizumab; these potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-08; Primary Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bevacizumab when administered concurrently with 5-fluorouracil (5-FU) and external beam radiation therapy (EBRT) in patients with cT3 and T4 rectal cancer prior to surgery | 29 days

SECONDARY OUTCOMES:
Pathological response rate after preoperative bevacizumab, 5-FU, EBRT, and surgery | Up to 5 years
Progression-free survival | From protocol entry until documented progression of disease or death from any cause, assessed up to 5 years
  The progression-free survival curve will be estimated using the Kaplan-Meier methods.
Local control | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Willett, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina